CLINICAL TRIAL: NCT02626897
Title: A Comparison of Two Wrist-worn Accelerometer Devices for the Measurement of Activity in Sarcoidosis Patients
Brief Title: A Comparison of Accelerometers for Measuring Daily Activity in Sarcoid
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of East Anglia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 1.3-27.11.2015
Record Dates: First submitted 2015-12-02; First posted 2015-12-10 (Estimated); Last update posted 2015-12-10 (Estimated); Status verified 2015-12

CONDITIONS: Sarcoidosis
Keywords: Sarcoidosis; Daily activity; Exercise; Accelerometer
MeSH Terms: conditions — Sarcoidosis; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sarcoidosis - GENEActiv device first (Other): Six patients start with the GENEActiv wrist-worn accelerometer which is needed to be worn for a 7 day period. Participants then switch to the ActiGraph GT3X device for a 7 day period. At the end of this second period they complete a short exit questionnaire detailing their experience and their device preference.
  Interventions: Device: GENEActiv Original Accelerometer; Device: ActiGraph GT3X Accelerometer
- Sarcoidosis - ActiGraph device first (Other): Six patients start with the ActiGraph GT3X wrist-worn accelerometer which is needed to be worn for a 7 day period. Participants then switch to the GENEActiv device for a 7 day period. At the end of this second period they complete a short exit questionnaire detailing their experience and their device preference.
  Interventions: Device: GENEActiv Original Accelerometer; Device: ActiGraph GT3X Accelerometer

INTERVENTIONS:
Device: GENEActiv Original Accelerometer — Wrist-worn device measuring accelerations as a measure of daily activity.
Device: ActiGraph GT3X Accelerometer — Wrist-worn device measuring accelerations as a measure of daily activity.

SUMMARY:
This cross-over study of 12 patients with sarcoidosis will look at two different widely-used accelerometer devices. These devices are wrist worn and similar in size to a wrist-watch. They measure daily activity levels. The investigators hope to use one of these devices in the future within a randomised-controlled trial looking at using methylphenidate for the treatment of sarcoidosis-associated fatigue. In order to ensure that the investigators choose the ideal device the investigators wish to compare the GENEActiv and ActiGraph GT3X devices. Participants will be required to wear the devices for 7 days each, with 6 patients beginning with the GENEActiv device and changing to the ActiGraph device after 7 days, the remaining 6 participants starting with the Actigraph before changing to the GENEActiv. Patients will complete a short exit questionnaire about their experience with the devices and their preference. The best device will be determined by both patient preference and reliability of collecting data.

DETAILED DESCRIPTION:
This will be a small comparator study comparing two devices (GENEActiv original and ActiGraph GT3X) in 12 patients with sarcoidosis. Participants wear one device for 7 days before returning the device, and wear the second device to wear for a further 7 day period. Each participant will wear the devices for 24 hours throughout the measurement period. The devices will be worn in a random order, randomised using sealed envelopes. They will be advised not to remove the devices during the 7 day monitoring period, with the exception of the GT3X which should be removed if the participant is bathing or swimming (they are able to shower). When each device is returned the participants will be asked to complete an exit questionnaire on their experience with the device. Before the participants wear the devices they will be asked to complete a short question regarding how tired/fatigued they feel.

The devices will be worn on the participant's non-dominant wrist. They will wear both devices in a random order (determined by randomisation at the start of the trial with regards to which device will be worn first). Six participants will start with the GENEActiv device and six will begin with the Actigraph GT3X device. The device order will be chosen randomly based upon a random number sequence generated in Microsoft Excel and placed in envelopes numbered 1 to 12.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female aged over 18
2. Diagnosed with sarcoidosis by either; biopsy confirming non-caseating granulomas consistent with sarcoidosis, or multi-disciplinary interstitial lung disease meeting diagnosis of sarcoidosis.
3. Ambulatory patient (not wheelchair or bed-bound)
4. Able to provide written informed consent

Exclusion Criteria:

1. Unable to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2016-01; Primary Completion 2016-03 (Estimated); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
Patient acceptability of devices | After 7 days of each device (day 7, day 14)
  Visual analogue scale measures of patient acceptability of devices

SECONDARY OUTCOMES:
Comparison of activity measures (time in moderate or vigorous activity) | After 7 days of each device (day 7, day 14)
  Comparison of time in moderate or vigorous activity between devices - is one device persistently recording lower levels of activity over the periods of activity?
Number of devices with valid data | After 7 days of each device (day 7, day 14)
  Number of devices recording minimum "valid" data (>10hrs day, 2 weekdays, 2 weekend days).
Number of devices with full data | After 7 days of each device (day 7, day 14)
  Number of devices recording "full" data (>16hrs/day, 7 days)

CONTACTS AND LOCATIONS:
Overall Officials: Chris Atkins, MB/BS, Principal Investigator — University of East Anglia; Andrew M Wilson, MD, Study Director — University of East Anglia
Locations (1):
- Norfolk and Norwich Univeristy Hospital NHS foundation Trust, Norwich, Norfolk, United Kingdom